CLINICAL TRIAL: NCT07107178
Title: A Phase Ib Study of the Safety, Tolerability and Efficacy of BT02 for the Treatment of Patients With Advanced Malignant Melanoma
Brief Title: A Clinical Study of BT02 for the Treatment of Patients With Advanced Malignant Melanoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biotroy Therapeutics (Industry)
Collaborators: Peking University Cancer Hospital and Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT02-102
Record Dates: First submitted 2025-07-16; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Advanced Melanoma; Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- dose escalation and expansion (Experimental)
  Interventions: Drug: BT02

INTERVENTIONS:
Drug: BT02 — monoclonal antibody injection with intravenous administration every 2 or 3 weeks

SUMMARY:
The goal of this clinical trial is to learn about the safety, tolerability and preliminary effectiveness of a treatment for patients with advanced melanoma,regardless of gender, aged between 18 and 75 years (inclusive).

Participants will receive the investigational product intravenously every two or three weeks. The treatment will continue for a maximum of two years for those who do not show signs of disease progression or experience intolerable side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed diagnosis of unresectable locally advanced or metastatic malignant melanoma (except for uveal melanoma) who have failed in the prior systemic therapy .
2. Adequate organ and hematologic function.
3. At least 1 extracranial measurable lesion.
4. An ECOG activity status score of 0-1.
5. A life expectancy of ≥ 3 months.
6. Eligible participants of childbearing potential (both males and females) must agree to using effective contraception throughout the study period.
7. Good compliance and willingness to follow up.

Exclusion Criteria:

1. Prior to first dose, received systemic antitumor therapy , scheduled major surgical procedure within 4 weeks , received systemic immunostimulants within 5 half-lives and systemic corticosteroids or other immunosuppressive medications within 14 days.
2. A history of active autoimmune disease within the past 2 years.
3. A history of clinically significant cardiovascular disease, severe cardiac rhythm/conduction abnormalities or LVEF<50%. A history of severe pulmonary disease that may lead to severe episodes of dyspnea.
4. A severe acute or chronic infection when enrollment.
5. Remaining the toxic reaction in previous anti-tumor therapy that has not recovered to ≤ Grade 1 .
6. Unresolved > grade 1 irAE or the history of a grade ≥ 3 irAE in previous immunotherapy, or known hypersensitivity to the formulation of the investigational product.
7. Clinically active CNS metastases or meningeal metastases.
8. A history of other type of malignancies.
9. Received a live attenuated vaccine within 28 days prior to the administration of the investigational product.
10. Poor compliance.
11. A history of alcohol/drugs abuse.
12. Current pregnancy or breastfeeding.
13. Other severe physical or mental illnesses or abnormal laboratory test results that the investigator deems unsuitable for participation in this study considering safety and compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Through the study completion, an average of 2 years
Dose limited toxicity(DLT) | Through the dose escalation phase, an average of 8 months
Maximum tolerable dose(MTD) | Through the dose escalation phase, an average of 8 months
Recommended phase 2 dose(RP2D) | Through the study completion, an average of 2 years

SECONDARY OUTCOMES:
Objective response rate (ORR) on tumor assessments | Through the study completion, an average of 2 years
Progression-free survival (PFS) on tumor assessments | Through the study completion, an average of 2 years
Overall survival (OS) | Through the study completion, an average of 2 years
Duration of response (DoR) on tumor assessments | Through the study completion, an average of 2 years
Disease control rate (DCR) on tumor assessments | Through the study completion, an average of 2 years
Mean and median Area under the curve (AUC) of BT02 following first dose and repeated administration at each dose level | Through the study completion, an average of 2 years
Mean and median Maximum concentration (Cmax) of BT02 following first dose and repeated administration at each dose level | Through the study completion, an average of 2 years
ADA and NAb incidence | Through the study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Undecided